CLINICAL TRIAL: NCT01018394
Title: A Pilot Study to Compare the Nicotine Lozenge and Tobacco-Free Snuff for Smokeless Tobacco Reduction
Brief Title: Nicotine Lozenge or Tobacco-Free Snuff for Smokeless Tobacco Reduction
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jon Ebbert, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-005172
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Results first posted 2013-09-13 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Tobacco Dependence
Keywords: tobacco dependence; tobacco reduction; chewing tobacco; snuff; moist snuff
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nicotine lozenges (Active Comparator): 40 subjects will be assigned to receive nicotine lozenges for 8 weeks. They will use the nicotine lozenges ad lib, up to 8 lozenges per day.
  Interventions: Drug: nicotine lozenges
- tobacco free snuff (Active Comparator): 41 subjects will receive tobacco free snuff for 8 -12 weeks. The tobacco-free snuff will be used ad lib - as needed.
  Interventions: Drug: tobacco-free snuff

INTERVENTIONS:
Drug: nicotine lozenges — 4 mg nicotine lozenges for a maximum duration of 12 weeks used ad lib - up to 8 nicotine lozenges per day.
  Arms: nicotine lozenges
Drug: tobacco-free snuff — Tobacco-free snuff used ad lib for a maximum of 12 weeks
  Arms: tobacco free snuff

SUMMARY:
Smokeless tobacco (ST) is a known human carcinogen. Long-term ST use is known to increase the risk for oropharyngeal cancer. Extant literature on cigarette smokers suggests that smoking reduction increases smoking abstinence among smokers not interested in quitting. The overarching goal of this line of research is to develop a ST reduction intervention among ST users not interested in quitting tobacco. Our first step is to conduct the proposed pilot study designed to assess the efficacy of the nicotine lozenges or tobacco-free snuff for reducing ST use or facilitating ST abstinence among ST users not interested in quitting.

DETAILED DESCRIPTION:
In this study, we will enroll 81 subjects who will be randomized to either the nicotine lozenge or tobacco-free snuff to reduce their ST use over 8 weeks with follow-up at 12 weeks. Forty subjects will be recruited at Mayo Clinic in Rochester, MN, and 40 subjects will be recruited at the Oregon Research Institute in Eugene, Oregon.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years of age;
2. no intention of quitting in the next one month;
3. report ST as their primary tobacco of use;
4. have used ST daily for the past 12 months;
5. have been provided with, understand, and have signed the informed consent
6. are able to complete all study visits;
7. are in general good health as determined by medical history.

Exclusion Criteria:

1. currently using or have used (within the past 30 days) any other behavioral or pharmacologic tobacco treatment program;
2. currently enrolled in another research study;
3. describe having a medical history of: (a) unstable angina; (b) myocardial infarction within the past 6 months; (c) cardiac dysrhythmia other than medication-controlled atrial fibrillation or paroxysmal supraventricular tachycardia; or (d) medically-treated or untreated hypertension with BP ≥ 180 systolic OR ≥ 100 diastolic;
4. have phenylketonuria (PKU) [nicotine lozenges contain aspartame which is metabolized to phenylalanine and not processed in individuals with PKU];
5. have another member of their household already participating in this study;
6. have other medical or psychiatric conditions that would exclude the participant in the opinion of the investigators;
7. have a score of ≥ 15 on the Patient Health Questionnaire (PHQ-8) on the phone call pre-screen;
8. are currently pregnant are trying to become pregnant;
9. are currently breast-feeding and unwilling to stop during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon O Ebbert, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Oregon Research Institute, Eugene, Oregon

REFERENCES:
- [Result] Ebbert JO, Severson HH, Croghan IT, Danaher BG, Schroeder DR. Comparative effectiveness of the nicotine lozenge and tobacco-free snuff for smokeless tobacco reduction. Addict Behav. 2013 May;38(5):2140-5. doi: 10.1016/j.addbeh.2013.01.023. Epub 2013 Feb 4. PMID 23454876

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on February 2010 and completed on September 2011. Interested subjects who passed a phone pre-screen were seen at a medical clinic (Mayo Clinic in Rochester, Minnesota and Oregon Research Institute in Eugene, Oregon) for consenting and additional study procedures to determine eligibility.
Groups:
- Nicotine Lozenges: Subjects will be assigned to receive nicotine lozenges for 8 weeks. They will use the nicotine lozenges ad lib, up to 8 lozenges per day.
  nicotine lozenges : 4 mg nicotine lozenges for a maximum duration of 12 weeks used ad lib - up to 8 nicotine lozenges per day.
- Tobacco Free Snuff: Subjects will receive tobacco free snuff for 8 -12 weeks. The tobacco-free snuff will be used ad lib - as needed.
  tobacco-free snuff : Tobacco-free snuff used ad lib for a maximum of 12 weeks
Period: Overall Study
Arm/Group | Nicotine Lozenges | Tobacco Free Snuff
Started | 40 | 41
Completed | 31 | 33
Not Completed | 9 | 8
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Lost to Follow-up | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine Lozenges | Tobacco Free Snuff | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 36 | 37 | 73
  >=65 years | 3 | 3 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 37.8 (15.9) | 37.5 (12.5) | 37.6 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 40 | 38 | 78
Baseline tobacco used per week [Mean (Standard Deviation); unit: cans of smokeless tobacco] — Amount of smokeless tobacco used upon study entry.
  cans of smokeless tobacco | 3.2 (2.1) | 4.0 (2.7) | 3.6 (2.4)

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Smokeless Tobacco Reduction Greater or Equal to 50%
Description: Percentage of participants who reduced smokeless tobacco use (cans per week) by 50% or more from baseline
Time Frame: baseline, week 4
Measure: Number; unit: percentage of participants
Arm/Group | Nicotine Lozenges | Tobacco Free Snuff
Number analyzed (Participants) | 40 | 41
percentage of participants | 25 | 19
Statistical Analysis 1: Comparison: Nicotine Lozenges vs Tobacco Free Snuff; The percentage of participants who reduced tobacco use by greater or equal to 50% from baseline was compared between groups using Fisher's exact test. A one tailed P of less than 0.2 was considered sufficient evidence to warrant a larger study; Test type: Superiority or Other; p = 0.108, Fisher Exact — A one tailed P of less than 0.2 was considered sufficient evidence to warrant a larger study; 1 tailed; Odds Ratio (OR) = 1.9, 95% CI 2-sided [0.7 to 5.1]

2. Primary Outcome: Tobacco Abstinence at 12 Weeks
Description: Number of participants who were biochemically confirmed abstinent from tobacco at week 12 using urinary anabasine less than 2 ng per ml.
Time Frame: week 12
Measure: Number; unit: participants
Arm/Group | Nicotine Lozenges | Tobacco Free Snuff
Number analyzed (Participants) | 40 | 41
participants | 8 | 5

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse Events were collected during the medication phase (baseline to week 12).
Arm/Group | Nicotine Lozenges | Tobacco Free Snuff
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 3/40 | 1/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nicotine Lozenges (N=40) | Tobacco Free Snuff (N=41)
sore throat (General disorders) | 1 | 1
dizziness (General disorders) | 1 | 0
insomnia (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes